CLINICAL TRIAL: NCT03923842
Title: Denosumab In Ebv Related Nasopharyngeal Carcinoma (Npc) As A Model For Rank-Mediated Immunologic Modulation Of Virus-Related Tumours - Dern Study
Brief Title: Denosumab In Ebv Nasopharyngeal Carcinoma As A Model For RankMediated Immunologic Modulation Of Virus-Related Tumours
Acronym: Dern
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Collaborators: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-005017-31
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Nasopharyngeal Carcinoma; EBV Related Carcinoma
Keywords: NPC; EBV
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: This is a phase II, 2:1 randomized, open label, and multicentre proof of principle trial with denosumab in patients with recurrent/metastatic (RM) NPC at first line systemic therapy.
Masking Description: NN
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A: Denosumab Treatment (Experimental): Denosumab 120 mg sc on day -15, -8 and day 1, followed by Denosumab 120 mg sc q4wks + platinum based drugs q3wks + Gemcitabine 1250 mg/sm day 1,8 q3wks for 6 cycles. Denosumab 120 mg sc q4wks will continue for 12 months since chemotherapy end.
  Interventions: Drug: Denosumab Inj 120 MG/1.7ML
- ARM B Control Arm (Active Comparator): platinum based drugs q3wks + Gemcitabine 1250 mg/sm day 1,8 q3wks for 6 cycles. At the end of the 6 cycles, if the patient is not progressing, can continue treatment with Gemcitabine alone.for 12 months
  Interventions: Drug: Chemotherapy as clinical standard of care

INTERVENTIONS:
Drug: Denosumab Inj 120 MG/1.7ML — Denosumab 120 mg sc on day -15, -8 and day 1, followed by Denosumab 120 mg sc q4wks + platinum based drugs q3wks + Gemcitabine 1250 mg/sm day 1,8 q3wks for 6 cycles. Denosumab 120 mg sc q4wks will continue for 12 months since chemotherapy end.
  Other Names: Denosumab treatment
  Arms: ARM A: Denosumab Treatment
Drug: Chemotherapy as clinical standard of care — platinum based drugs q3wks + Gemcitabine 1250 mg/sm day 1,8 q3wks for 6 cycles. Gemcitabine will continue for 12 months if the patient will not shown disease progression
  Other Names: Standard of care treatment
  Arms: ARM B Control Arm

SUMMARY:
The aim of the present investigation is to test of the modulation obtained with denosumab as "priming" therapy before the start of chemotherapy and as concurrent therapy in a population of first line NPC recurrent/metastatic patients

DETAILED DESCRIPTION:
Approximately 15-20% of the cancers recognize infectious agents as causal factors. Epstein Barr Virus (EBV) is considered carcinogenic to humans for haematological and solid neoplasms such as nasopharyngeal carcinoma (NPC). Oncogenic mechanisms linking EBV with NPC need to be better delineated. However, the well-defined patterns of EBV cancer cells infection, together with its encoded regulated genes in tumours offers an option for immunological therapeutic strategies.

Distant metastases, especially of the bone, occurs in up to half of patients with NPC. This underlines the importance of improving systemic disease control.

Intravenous bisphosphonates (BP) are effective treatments for skeletal-related events (SRE) in patients with bone metastases. BPs also showed antitumor properties in solid malignancies by inhibiting cancer cell proliferation, inducing apoptosis and affecting bone microenvironment, increasing progression free survival (PFS) and overall survival (OS).

In head and neck squamous cell cancer, RANKL expression has been observed and correlated with tumour differentiation and progression. RANKL expression is also found in tumour-infiltrating Tregs. Once expressed, RANKL regulates epidermal dendritic cells and increases the number of Tregs, thereby suppressing excessive response to environmental stimuli. In NPC, the role of Tregs has been described and implicated in EBV-associated carcinogenesis.

Although no direct evidence of denosumab activity in NPC cells are available, its target's effect on Tregs is at the base of an indirect effect to tackle cancer immune evasion. In this scenario, treatment with RANK and RANKL inhibitors will supposedly act as positive immunoregulator reducing bone events but also improving treatment effects.

RANK expression was confirmed on 17 metastatic relapses of NPC treated at Fondazione IRCCS Istituto Nazionale dei Tumori, Milano.

The recent introduction of denosumab, a new drug active on bone metastases, with a different mechanism of action compared to BPs, changed the scenario. Denosumab is a fully human monoclonal antibody preventing the binding of RANKL to its receptor on osteoclasts' membrane. Denosumab is formulated for SC injection and for oncology indications is administered at a dose of 120 mg Q4W. Denosumab (120 mg SC) is approved worldwide for the prevention of SREs in patients with bone metastases from solid tumors and for the treatment of adults and skeletally mature adolescents with GCTB.

The above premises warrant the investigation of the activity of denosumab - an antibody competing with RANK, enhancing increasing tumour-specific immunity through the blockade of RANKL-regulated Tregs.

ELIGIBILITY:
Inclusion Criteria:

1. EBV related nasopharyngeal cancer
2. Detectable and quantifiable plasmatic EBV DNA
3. Recurrent and/or metastatic disease not suitable for curative treatment
4. PS < 2
5. Suitable for polychemotherapy
6. Age ≥ 18 years
7. Informed consent signed
8. Subject has adequate organ functions, evidenced by the following:

   1. AST (SGOT), ALT (SGPT) ≤ 2.5 x upper limit of normal range (ULN), or ≤ 5 x ULN range if liver metastasis present
   2. Total bilirubin ≤ 1.5 x ULN
   3. creatinine clearance 24/h > 50 mL/min
   4. Total serum calcium > 8.8 mg/dL
   5. Absolute neutrophil count ≥ 1.5 x 10*9 cells/L
   6. Platelets ≥ 100 x 10*9 cells/L
   7. Haemoglobin ≥ 9 g/dL
9. If of childbearing potential, willingness to use effective contraceptive method (Pearl Index < 1; e.g. oral contraceptive (pill), hormone spiral, hormone implant, transdermal patch, a combination of two barrier methods (condom and diaphragm), sterilisation, sexual abstinence) for the study duration and 5 months post-dosing.
10. Subject understands and voluntarily signs an ICF prior to any study-related assessments/procedures are conducted.
11. Subject is able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

1. Having received 1 or more chemotherapy line for recurrent/metastatic disease
2. Any residual CTCAE grade ≥ 2 toxicity
3. Subject has any other malignancy within 3 years prior to randomization, with the exception of adequately treated in situ carcinoma of the cervix, uteri, or non-melanoma skin cancer (all treatment of which should have been completed 6 months prior to enrolment), in situ squamous cell carcinoma of the breast, or incidental prostate cancer T1a, Gleason < 7, PSA <10 ng/ml.
4. Subject has had radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting IP, and/or from whom ≥ 30% of the bone marrow was irradiated.
5. Having participated in another clinical trial or having received any investigational agent in the preceding 30 days before study entry.
6. Chronic systemic immunosuppressive therapy that cannot be interrupted during treatment study.
7. Subject has significant active cardiac disease within the previous 6 months including unstable angina or angina requiring surgical or medical intervention, significant cardiac arrhythmia, or New York Heart Association (NYHA) class 3 or 4 congestive heart failure.
8. Subject has a known or suspected hypersensitivity to study drugs.
9. Subject is pregnant or breast feeding.
10. Subject is receiving prohibited medication as per section 7.4.2 and suspension of such treatment is considered unsafe.
11. Subject has history of prior or current osteonecrosis of the jaw (ONJ).
12. Subject has history of prior irradiation to the mandible, specified as:

    Dose constraints to the mandible: Dmax = 70 Gy, V50 = 62 Gy and V60 = 20 Gy Mandible should be contoured as whole organ, with alveolar bone, excluding teeth
13. Subject has any other concurrent severe and/or uncontrolled medical condition that would, in the Investigator's judgment, contraindicate subject participation in the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-06-30 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
plasmatic EBV DNA change | change in circulating EBV DNA levels from baseline (prior to the first denosumab administration on day -15 with respect to first chemotherapy administration
  Meaningful plasmatic EBV DNA change in circulating EBV DNA levels from baseline (prior to the first denosumab administration on day -15 with respect to first chemotherapy administration) to the third denosumab dose (denosumab day 16, equivalent to chemotherapy treatment day 1).

SECONDARY OUTCOMES:
Progression Free Survival | PFS will be defined as the time from Chemotherapy treatment start (day1 for chemotherapy, day16 for denosumab) to disease progression or death from any cause.
  PFS in patients treated or not with denosumab

OTHER OUTCOMES:
Absolute change in cellular immunity to EBV | prior to first denosumab administration, chemotherapy day -15 and denosumab day 1) and the subsequent planned time point (16 days, 2 and 6 months after denosumab treatment start
  Cellular immunity will be defined blood lymphocytes activity against LMP and EBNA antigens. Absolute change will be defined as the difference in such activity from baseline (i.e. prior to first denosumab administration, chemotherapy day -15 and denosumab day 1) and the subsequent planned time point (16 days, 2 and 6 months after denosumab treatment start).
Safety profile of denosumab plus chemotherapy: NCI CTCAE v 4.03 | During study treatment anf follow up period
  type and frequency of treatment-emergent adverse events, graded according to NCI CTCAE v 4.03
Absolute change in blood and salivary miRNA NPC profiles | at 16 days, 2 and 6 months after Denosumab treatment start
  (chosen among selected miRNAs having previously shown correlation with immune activity and with NPC), measured at each planned time point (at 16 days, 2 and 6 months after Denosumab treatment start
Absolute change of serum levels of RANKL and its inhibitor osteoprotegerin | at 16 days, 2 and 6 months after treatment start
  Absolute change of serum levels of RANKL and its inhibitor osteoprotegerin (OPG), measured at each planned time point
Absolute change in EBV DNA levels at each other planned time point | at 2 months after denosumab treatment start, prior to administration of 3rd denosumab treatment, and at 6 months, prior to administration of 7th denosumab treatment
  change in EBV DNA levels

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bossi, Dr., Study Chair — Università degli Studi di Brescia ASST degli Spedali Civili di Brescia
Locations (2):
- Italy (2):
  - ASST degli Spedali Civili di Brescia, Brescia
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan

IPD SHARING:
Plan to Share IPD: Undecided